CLINICAL TRIAL: NCT06647511
Title: Digital Solutions to Reduce Maternal Morbidity and Mortality in Pregnant Refugee Women
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Academy of Medicine (Unknown); Cornell University (Other); Apple Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-01026913
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Gestational Hypertension
Keywords: refugee; pregnant; digital
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Refugees: Participants will complete validated questionnaires, regular blood pressure measurements, pain and trauma assessments, and clinical monitoring during this study.
  Interventions: Device: Nokia-Withings BPM Connect Blood Pressure Monitor; Device: Smartwatch Devices

INTERVENTIONS:
Device: Nokia-Withings BPM Connect Blood Pressure Monitor — At-home blood pressure (BP) measurements will be weekly via a blood pressure cuff (e.g., Nokia-Withings BPM (Beats per Minute) Connect), with measurements being manually entered into the study specific smartphone app.
Device: Smartwatch Devices — Passive continuous collection of digital data (e.g., daily heart rate trends, activity levels, sleep measurements) for exploratory outcomes will occur via Apple Watches and Fitbit Versa 3s, which are synced to a smartphone application.

SUMMARY:
The goal of this observational study is to use digital health tracking to improve how high blood pressure and other health issues are detected in pregnant refugee women. The main questions this study aims to answer are are:

* Can a digital monitoring system that checks for high blood pressure in these women be tested and refined, using clinical training and validation?
* Can this digital monitoring system accurately track any related pregnancy health issues and be used to refer participants to care providers?
* Can this system be used to accurately identify risks associated with the contraction of pregnancy-related conditions, such as preeclampsia and high blood pressure?

Participants will:

* Complete baseline and follow-up in-person appointments;
* Complete surveys at these appointment that track their health, stress levels, and comorbidities/risks associated with pregnancy;
* Be given a smartwatch fitness tracker and electronic blood pressure cuffs for at-home measurements.

DETAILED DESCRIPTION:
The objective of this application, funded by the National Academy of Medicine Catalyst Award, is to maximize the performance of a digital cardiovascular monitoring system to detect gestational hypertension in pregnant refugee women. The central hypothesis is that the application of these digital health technologies will be able to diagnose gestational hypertension in refugee mothers with 85% sensitivity as compared to the gold standard (clinical diagnosis). The rationale for this investigation is to improve the diagnosis of hypertension in refugee mothers, leading to targeted treatment.

This study's primary objective is to maximize the performance of digital health monitoring systems to detect gestational hypertension through system training and validation. The investigators aim to do this by utilizing technologies such as smartwatches and electronic blood pressure monitors to track health data throughout enrollment. Tracking this health data will also allow study investigators to track several other comorbid conditions in refugee mothers. This collection will take place over 24 months to train and validate this digital system. The performance of the prediction models will be assessed using two measures: Receiver Operating Characteristic (ROC) curve analysis, which evaluates the model's discrimination ability between disease states; and the Integrated Brier Score (cumulative mean squared error over time) will provide data on the model's predictive accuracy and reliability.

The secondary objectives of this study are to document comorbid illness and stress, assess the program's ability to make successful referrals, and connect the study population with healthcare providers for primary care visits. This will be completed by digital health tracking and the retention of contact with the participants throughout the duration of their enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Refugee, asylum seeking, or asylee as designated by the U.S. Government
* Greater than or equal to 18 years of age
* Has a personal smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Determined by the PI to be in an extremely vulnerable position and therefore not suited for research participation
* Planned move from the New York City (NYC) area within the next 24 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is a pregnant refugee, or asylee as designated by the U.S. Government.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Digital Sensitivity for detecting gestational hypertension (HTN) | 13 months [maximum duration of enrollment]
  The diagnostic accuracy of the digital blood pressure cuffs will be compared to the measurements taken during in-person visits.

SECONDARY OUTCOMES:
Number of Participants that Complete All Surveys Between Appointments | 13 months [maximum duration of enrollment]
  The completion of weekly surveys will be assessed for each participant and the number of participants that complete all surveys sent to them will be compared to the overall number of participants enrolled.
Number of Participants That Complete All Surveys at the Baseline Appointment | 13 months [maximum duration of enrollment]
  The number of participants that complete every single survey at the baseline appointment out of the total number of participants will be recorded.
Number of Participants Referred to Physicians/Care that do not have a designated provider | 13 months [maximum duration of enrollment]
  Participants without designated care providers during their pregnancy will be noted and the number of participants that are successfully referred to physicians/other providers will be recorded.
Number of Participants With No Comorbid Pain as Assessed by BPI-SF | 13 months [maximum duration of enrollment]
  Chronic pain will be evaluated using the validated Brief Pain Inventory - Short Form (BPI-SF). The mean BPI-SF score quantifies pain severity (worst, least, average, and now) and pain interference into the following: none (score 0), mild (1-4), moderate (4-6), or severe (7-10).The number of participants who score 0 on the BPI-SF will be measured.
Number of Participants With Mild Comorbid Pain as Assessed by BPI-SF | 13 months [maximum duration of enrollment]
  Chronic pain will be evaluated using the validated Brief Pain Inventory - Short Form (BPI-SF). The mean BPI-SF score quantifies pain severity (worst, least, average, and now) and pain interference into the following: none (score 0), mild (1-4), moderate (4-6), or severe (7-10).The number of participants who score from 1-4 on the BPI-SF will be measured.
Number of Participants With Moderate Comorbid Pain as Assessed by BPI-SF | 13 months [maximum duration of enrollment]
  Chronic pain will be evaluated using the validated Brief Pain Inventory - Short Form (BPI-SF). The mean BPI-SF score quantifies pain severity (worst, least, average, and now) and pain interference into the following: none (score 0), mild (1-4), moderate (4-6), or severe (7-10).The number of participants who score from 4-6 on the BPI-SF will be measured.
Number of Participants With Severe Comorbid Pain as Assessed by BPI-SF | 13 months [maximum duration of enrollment]
  Chronic pain will be evaluated using the validated Brief Pain Inventory - Short Form (BPI-SF). The mean BPI-SF score quantifies pain severity (worst, least, average, and now) and pain interference into the following: none (score 0), mild (1-4), moderate (4-6), or severe (7-10).The number of participants who score from 7-10 on the BPI-SF will be measured.
Number of Participants with Low Comorbid Stress as Assessed by the PSS | 13 months [maximum duration of enrollment]
  Stress levels will be evaluated using the validated Perceived Stress Scale (PSS). The PSS ranges from 0 to 40, with 0-13 considered low stress, 14-26 considered moderate stress, and 27-40 considered high stress. The number of participants who score from 0-13 will be measured.
Number of Participants with Moderate Comorbid Stress as Assessed by the PSS | 13 months [maximum duration of enrollment]
  Stress levels will be evaluated using the validated Perceived Stress Scale (PSS). The PSS ranges from 0 to 40, with 0-13 considered low stress, 14-26 considered moderate stress, and 27-40 considered high stress. The number of participants who score from 14-26 will be measured.
Number of Participants with High Comorbid Stress as Assessed by the PSS | 13 months [maximum duration of enrollment]
  Stress levels will be evaluated using the validated Perceived Stress Scale (PSS). The PSS ranges from 0 to 40, with 0-13 considered low stress, 14-26 considered moderate stress, and 27-40 considered high stress. The number of participants who score from 27-40 will be measured.
Number of Participants with Comorbid Stress as Assessed by the SOIS | 13 months [maximum duration of enrollment]
  Stress levels will be evaluated using the validated Stress of Immigration Survey (SOIS). The SOIS is considered positive if any item on the survey is "yes," with the mean of all items giving an overall severity score from 1-5.
Number of Participants Who Score Positive for PTSD Symptoms on the HTQ | 13 months [maximum duration of enrollment]
  Mental health status will be evaluated using the validated Harvard Trauma Questionnaire (HTQ). The HTQ is positive for PTSD symptoms if the average score from Part IV is ≥2.5. The number of participants who have a positive score on the HTQ will be recorded.
Number of Participants Who Score Positive for Anxiety on the HSCL | 13 months [maximum duration of enrollment]
  Mental health status will be evaluated using the Hopkins Symptoms Checklist (HSCL). the HSCL is positive for anxiety if the average of items 1-10 or total averaged score is more than or equal to 1.75. The number of participants who have a positive score on the HSCL for anxiety will be recorded.
Number of Participants Who Score Positive for Depression on the HSCL | 13 months [maximum duration of enrollment]
  Mental health status will be evaluated using the Hopkins Symptoms Checklist (HSCL). the HSCL is positive for depression if the average of items 11-25 or total averaged score is more than or equal to 1.75. The number of participants who have a positive score on the HSCL for depression will be recorded.
Number of Participants with Cardiovascular Risk Factors and Disease as Assessed by the WHO Rose Angina Questionnaire. | 13 months [maximum duration of enrollment]
  Participants will be assessed for cardiovascular risk factors and disease using the World Health Organization (Rose) Angina Questionnaire (WHOAQ). The WHOAQ is deemed positive if any symptoms are recorded on the survey.
Number of Participants with Low Cardiovascular Risk Factors and Disease as Assessed by the AHA Atherosclerotic Cardiovascular Disease Pooled Cohort Equation | 13 months [maximum duration of enrollment]
  Cardiovascular risk factors and disease will be assessed using the American Heart Association (AHA) atherosclerotic cardiovascular disease (ASCVD) Pooled Cohort Equation (PCE) risk estimator. AHA ASCVD PCE Scores identify the risk of first occurrence of myocardial infarction or stroke. A score of less than 5% is low; 5%-7.5% is borderline; 7.5%-20% is intermediate; ≥20% is high. The number of participants that score less than 5% will be measured.
Number of Participants with Borderline Cardiovascular Risk Factors and Disease as Assessed by the AHA Atherosclerotic Cardiovascular Disease Pooled Cohort Equation | 13 months [maximum duration of enrollment]
  Cardiovascular risk factors and disease will be assessed using the American Heart Association (AHA) atherosclerotic cardiovascular disease (ASCVD) Pooled Cohort Equation (PCE) risk estimator. AHA ASCVD PCE Scores identify the risk of first occurrence of myocardial infarction or stroke. A score of less than 5% is low; 5%-7.5% is borderline; 7.5%-20% is intermediate; ≥20% is high. The number of participants who score from 5%-7.5% will be measured.
Number of Participants with Intermediate Cardiovascular Risk Factors and Disease as Assessed by the AHA Atherosclerotic Cardiovascular Disease Pooled Cohort Equation | 13 months [maximum duration of enrollment]
  Cardiovascular risk factors and disease will be assessed using the American Heart Association (AHA) atherosclerotic cardiovascular disease (ASCVD) Pooled Cohort Equation (PCE) risk estimator. AHA ASCVD PCE Scores identify the risk of first occurrence of myocardial infarction or stroke. A score of less than 5% is low; 5%-7.5% is borderline; 7.5%-20% is intermediate; ≥20% is high. The number of participants who score from 7.5%-20% will be measured.
Number of Participants with High Cardiovascular Risk Factors and Disease as Assessed by the AHA Atherosclerotic Cardiovascular Disease Pooled Cohort Equation | 13 months [maximum duration of enrollment]
  Cardiovascular risk factors and disease will be assessed using the American Heart Association (AHA) atherosclerotic cardiovascular disease (ASCVD) Pooled Cohort Equation (PCE) risk estimator. AHA ASCVD PCE Scores identify the risk of first occurrence of myocardial infarction or stroke. A score of less than 5% is low; 5%-7.5% is borderline; 7.5%-20% is intermediate; ≥20% is high. The number of participants who score above 20% will be measured.
Number of Participants with Cardiovascular Risk Factors and Disease as Assessed by the QVSFS | 13 months [maximum duration of enrollment]
  Participants will be assessed for cardiovascular risk factors and disease by using the Questionnaire for Verifying Stroke-Free Status (QVSFS). The QVSFS is positive if any questions are answered in the affirmative.

CONTACTS AND LOCATIONS:
Overall Officials: Gunisha Kaur, MA, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No